CLINICAL TRIAL: NCT00405561
Title: A Prospective, Open, Single-Arm, Multicenter Phase II Clinical Trial to Evaluate the Progression Free Survival and Safety in Patients With Advanced Colorectal Carcinoma Treated With AMT2003
Brief Title: Study to Evaluate Progression Free Survival in Cancer Patients With Advanced Colorectal Carcinoma With AMT2003
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Auron Healthcare GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMT/P2GI/001 Part III; LC001Auron2005
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Colorectal Carcinoma
Keywords: Advanced Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms

ARMS (1):
- AMT2003 (Experimental)
  Interventions: Drug: AMT2003

INTERVENTIONS:
Drug: AMT2003

SUMMARY:
The purpose of the study is to evaluate efficacy and safety of AMT2003 in cancer patients with advanced colorectal carcinoma.

The primary endpoint is progression free survival rate at 18 weeks after registration

DETAILED DESCRIPTION:
The study will include patients with advanced colorectal carcinoma that is refractory to standard therapy or for which no effective standard therapy exists. Eligible patients must have had at least second-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Cancer confirmed by histology or cytology
* At least one measurable lesion
* Advanced disease refractory to standard therapy or for which no standard therapy exists
* Life expectancy of at least 3 months

Exclusion Criteria:

* Known secondary neoplasia or central nervous system (CNS) metastases; acute or chronic leukemia, lymphoma or multiple myeloma
* Body weight below 45 kg
* Female patients who are pregnant or breast feeding or adults of reproductive potential not employing effective method of birth control
* Confirmed diagnosis of HIV
* Insulin dependent diabetes mellitus / abnormal glucose tolerance test (GTT) / latent diabetes mellitus type I or II
* Chemotherapy or radiotherapy less than 4 weeks prior to entry
* Surgery less than 2 weeks prior to entry (or not recovered from effects of surgery)
* Participation in a clinical trial less than 30 days prior to entry in the study

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2006-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival;at 18 weeks after registration | 2010

SECONDARY OUTCOMES:
Best overall response rate (ORR, CR and PR) within 18 weeks after registration | 2010
Progression Free survival time (PFS), over complete observation period | 2010
Overall Survival (OS) time | 2010
Quality of Life (EORTC QLQ-C30) and Performance Status (Karnofsky Index) | 2010
Safety and Tolerability | 2010

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Drevs, PD Dr. med., Principal Investigator — Clinic Sanafontis, Freiburg
Locations (1):
- Clinic SanaFontis, Freiburg im Breisgau, Germany

REFERENCES:
- See also: now legally responsible for this study — http://www.alpiniainstitute.com